CLINICAL TRIAL: NCT03634436
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability Study Following A Single Subcutaneous Injection of SHR-1209 in Healthy Subjects
Brief Title: The PK/PD Study of A Single Subcutaneous Injection of SHR-1209 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1209-101
Record Dates: First submitted 2018-08-06; First posted 2018-08-16 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2019-09

CONDITIONS: Hypercholesteremia
Keywords: SHR-1209 Phase 1
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): A single subcutaneous injection of SHR-1209 dose 1 versus placebo
  Interventions: Drug: SHR-1209; Drug: Placebo
- Cohort 2 (Experimental): A single subcutaneous injection of SHR-1209 dose 2 versus placebo
  Interventions: Drug: SHR-1209; Drug: Placebo
- Cohort 3 (Experimental): A single subcutaneous injection of SHR-1209 dose 3 versus placebo
  Interventions: Drug: SHR-1209; Drug: Placebo
- Cohort 4 (Experimental): A single subcutaneous injection of SHR-1209 dose 4 versus placebo
  Interventions: Drug: SHR-1209; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1209 — Pharmaceutical form: lyophilized formulation
  Route of administration: subcutaneous
Drug: Placebo — Pharmaceutical form: lyophilized formulation
  Route of administration: subcutaneous

SUMMARY:
This is a Single Center, Randomized, Double-blind, Dose Escalation, Placebo Parallel Controlled PhaseⅠClinical study to Evaluate the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics with A Single Subcutaneous Injection of SHR-1209 in Healthy Subjects.

The primary objective of this study is to investigate the safety and tolerability of a range of subcutaneous SHR-1209 in healthy subjects. Secondary objectives are to determine the pharmacokinetics (PK) and pharmacodynamics(PD) profile of SHR-1209 in healthy subjects including assessment of immunogenicity.

DETAILED DESCRIPTION:
32 adult healthy subjects with 4 dose groups will be enrolled in the study, including two subjects in the lowest dose group, all of whom received the SHR-1209 without placebo control. The other three groups have 10 subjects in each group, 8 administered SHR-1209 and 2 administered placebo. The primary endpoint is the Safety and Tolerability : adverse events, vital signs, physical examination, laboratory examination, 12 lead electrocardiogram, injection site reactions, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤45 years old;
2. The body mass index (BMI) should be 19 or greater and < 28kg/m2, the male weigh ≥50.0kg and <90.0kg, and the female weigh ≥45.0kg and <90.0kg;
3. Serum LDL-C concentration≥2.0mmol/L and < 4.1mmol/L;
4. Fasting triglycerides < 2.3 mmol/L;
5. The comprehensive physical examination is eligible or slightly abnormal but the researchers determine no clinical implication.
6. Signed informed consent.

Exclusion Criteria:

1. Subjects determined by the researchers have diseases that affect drug absorption, distribution, metabolism and excretion or low compliance;
2. A clinical history of drug allergy or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known allergy to experimental or similar experimental drugs;
3. Serum creatinine exceeded the upper limit of normal value (ULN) during screening;
4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma pancreatic acyl transferase (GGT), more than 2 x ULN, or total bilirubin more than 1.5 x ULN during screening;
5. Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) were positive;
6. Subjects with previous malignant tumor diseases;
7. 3 months prior to screening involved in any drug or medical device clinical subjects, or within 5 half-life of drugs (test drug half-life more than 3 months) before screening. etc

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Pre-dose to 150 days after dose administration

SECONDARY OUTCOMES:
Assessment of PK parameter-time to maximum concentration (Tmax) | Pre-dose to 150 days after dose administration
Assessment of PK parameter-maximum concentration (Cmax) | Pre-dose to 150 days after dose administration
Assessment of PK parameter-area under curve (AUC) | Pre-dose to 150 days after dose administration
Assessment of PD parameter-change in Low-Density Lipoprotein Cholesterol (LDL-C) from baseline | Pre-dose to 150 days after dose administration
Assessment of PD parameter-change in Total Cholesterol (T-C) from baseline | Pre-dose to 150 days after dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- FuWai Hospital , Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053